CLINICAL TRIAL: NCT03968536
Title: Measuring the Impact of a Multimodal Intervention on Falls and Fear Falls Among People 65 Years Old, Residents at Home
Acronym: KitPA
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02910-55
Record Dates: First submitted 2019-02-20; First posted 2019-05-30 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Fall; Old Age; Atrophy
MeSH Terms: conditions — Atrophy | interventions — Ergonomics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: fall prevention — Training in physiotherapy sessions and ergonomic home development
  Other Names: ergonomics

SUMMARY:
Measuring the Impact of a Multimodal Intervention on Falls and Fear Falls among People 65 Years Old, Residents at Home in Boulogne city

DETAILED DESCRIPTION:
We hypothesize that participation in the multimodal program " Autonomy Prevention Kit " would lead to a decrease in falls and the fear of falling.

this study targets retired people, 65 years of age and over, living at home, identified as being independent (Iso Group Resources type 4-5-6 without formal validation being carried out) but who represent statistically an increased risk of falls in comparison to the general population.

The inclusion takes place before the first session of the Equilibr'Age® workshop. Subjects will have already benefited from a first collective information organized by the Boulogne City Council (see annexes of the CRF). 3 times mark the collection of data.

At the time of inclusion, at the end of the 12 sessions of the Equilbr'Age® workshop (M3) and 3 months after the end of the workshop ( 6 months after the beginning of inclusion).

The study does not involve new acts since it is only an assessment of the effects of a protocol that proposes non-sports activities as well as advice to citizens of the municipality.

ELIGIBILITY:
Inclusion Criteria:

* Retired
* Age ≥ 65 years;
* GIR ≥ 4
* Commitment to participate in all interventions of the "autonomy prevention" Kit
* Autonomous in its travels
* The person expressed no objection to participating in the KitPA study.

Exclusion Criteria:

* In professional activity
* Age < 65 years;
* GIR < 4
* Person under guardianship or curatorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Autonomous elderly people walking
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the number of falls before/after and the fear of falling before/after according Equilibr'Age® workshop | 6 months
  Equilibr'Age® workshop

SECONDARY OUTCOMES:
Comparison of life quality before/after according EQ-ED scale | 6 months
  Quality of life scale

OTHER OUTCOMES:
Assesssment of health status according Self Perceived Health (SPH) scale | 6 months
  Self Perceived Health (SPH) scale
Assessment of the impacte of workshops according Likert scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Nicolas, master, Principal Investigator — Gérond'if
Locations (1):
- Gerond'if, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No